CLINICAL TRIAL: NCT03243331
Title: An Initial Safety Study of Gedatolisib Plus PTK7-ADC for Metastatic Triple-negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kathy Miller (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0613
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Triple Negative Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — gedatolisib; cofetuzumab pelidotin

STUDY DESIGN:
Intervention Model Description: Study will enroll 3 patients to the cohort 1 dose level. If 0 of 3 patients experience a DLT, the study will proceed to cohort 2. If 1 patient experiences a DLT, 3 additional patients will be enrolled into cohort 1. If 1 of 6 patients experience a DLT, the study will proceed and 3 patients will be enrolled to the cohort 2 dose level. If 0 patients experience a DLT in cohort 2, the study will proceed to cohort 3. If 1 patient experiences a DLT at cohort 2, 3 additional patients will be enrolled into cohort 2. If the study proceeds to cohort 3, 3 patients will be enrolled at this dose level. If 0 patients experience a DLT, the study will enroll an additional 3 patients at the cohort 3 dose level to better define the safety profile. If 1 of 3 patients experiences a DLT at cohort 3, 3 additional patients will still be enrolled into cohort 3. If 1 of 6 patients experience a DLT, the study will complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gedatolisb + PTK7-ADC (Experimental)
  Interventions: Drug: Gedatolisib; Drug: PTK7-ADC

INTERVENTIONS:
Drug: Gedatolisib — Gedatolisb will be intravenously administered on Day 1, Day 8 and Day 15 of every 21 day cycle at a dose of 110 mg or 180mg depending on cohort assignment.
Drug: PTK7-ADC — PTK7-ADC will be administered on Day 1 of every 21 day cycle at a dose of 1.4mg/kg or 2.8 mg/kg depending on cohort assignment.
  Other Names: PF-06647020

SUMMARY:
Phase 1 study to evaluate the safety and effect of Gedatolisib and PTK7-ADC for the treatment of triple negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Triple-negative Breast Cancer
* Willingness to undergo tumor biopsy
* Patients must have received at least 1 prior chemotherapy regimen for metastatic disease

Exclusion Criteria:

* Previous treatment with mTOR inhibitor
* Untreated brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Safety of Gedatolisb + PTK7-ADC using NCI CTCAE v4.0 | through study completion i.e. up to 1 year
  safety and toxicity data will be assessed using NCI CTCAE v4.0 and tabulated and reported

SECONDARY OUTCOMES:
Efficacy in all enrolled subjects | 18 weeks
  efficacy as determined by clinical benefit at 18 weeks
Overall response rate in all enrolled subjects | through study completion i.e. up to 1 year
  efficacy as determined by overall response rate
Progression free survival in all enrolled subjects | through study completion i.e. up to 1 year
  efficacy as determined by progression free survival
Pharmacodynamic determination of inhibition of PI3k signaling | Cycle 1 Day 15
  Pathological H-score will be determined from tissue obtained at screening and Cycle 1 Day 15. H-score will be compared to calculate percentage inhibition between samples.
Pharmacodynamic determination modulation of Wnt pathway | Cycle 1 Day 15
  pathological H-score will be determined from tissue obtained at screening and Cycle 1 Day 15. H-score will be compared to calculate percentage change in expression between samples.
Pharmacodynamic determination modulation of Wnt pathway | Cycle 1 Day 15
  RNA sequencing of tissue collected at screening and Cycle 1 Day 1 to compare Wnt pathway expression after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University; Milan Radovich, PhD, Principal Investigator — Indiana University
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States